CLINICAL TRIAL: NCT05476744
Title: Viral Clearance and Epidemiological Characteristics in Patients With Monkeypox
Acronym: MoViE
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other); CEEISCAT (Unknown)
Responsible Party: Principal Investigator, Oriol Mitja, Associate Professor, Infectious Diseases and Global Heaelth, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Other Study IDs: MoViE Study
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Monkeypox
Keywords: Monkeypox; Viral clearance; Viral dynamics
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Skin lesions, blood, throat, rectum, semen, and vaginal fluid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present observational study has been designed to understand the dynamics of viral clearance amongst patients with confirmed monkeypox, by quantifying monkeypox viral load in different specimens trough time, to better inform decision-making about patient management and isolation guidelines. Also, an immune analysis will be performed in a subset of individuals to describe humoral and cellular responses to monkeypox.

DETAILED DESCRIPTION:
Starting in early May 2022 a large number of cases of Monkeypox have been reported in non-endemic countries. Although initial cases appeared to be linked to travel, the majority of subsequent cases appear to have no travel associated risk factors and these cases have predominantly occurred amongst Men who have Sex with Men (MSM) suggesting autochthonous transmission associated with sexual networks.

Monkeypox is known to be transmitted by close contact with skin lesions of infected individuals and/or via droplets. It is known that the virus can be detected from skin lesions, in blood, in throat swabs and on occasion urine samples. There is limited information as to whether the virus can be detected or persist in other sites including semen. Serial virological monitoring has been conducted in a small number of individuals and demonstrates that prolonged shedding for at least 2-3 weeks appears to be relatively common. To help control the current outbreak health authorities have used a number of strategies including identifying and isolating cases of monkeypox combined with contact tracing and limited use of ring-vaccination strategies. Because the number of cases seen outside of endemic areas has previously been limited, there is inadequate data to guide decision-making about the duration of isolation, but this is critical to the management of the current outbreak.

The present observational study has been designed to understand the dynamics of viral clearance amongst patients with confirmed monkeypox, by quantifying monkeypox viral load in different specimens trough time, to better inform decision-making about patient management and isolation guidelines. Also, an immune analysis will be performed in a subset of individuals to describe humoral and cellular responses to monkeypox.

ELIGIBILITY:
* Inclusion Criteria

  1. Adult male or female individuals of ≥18 years old.
  2. Examined by a specialist in sexually transmitted infections (STIs) and found to have lesions suggestive of monkeypox.
  3. Symptomatic with symptoms onset date ≤10 days prior to screening/baseline visit.
  4. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the trial.
  5. Has understood the information provided and capable of giving informed consent.
* Exclusion criteria:

  1. Severe disease - defined as requires admission to hospital
  2. Inability to consent and/or comply with trial protocol
  3. An alternative confirmed diagnosis that can fully explain the illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with monkeypox infection.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Viral clearance in skin lesions | From day 1 to day 57
  Time to undetectable monkeypox viral load in skin lesions (Number of days)
Viral clearance in blood | From day 1 to day 57
  Time to undetectable monkeypox viral load in blood (Number of days)
Viral clearance in oropharyngeal swabs | From day 1 to day 57
  Time to undetectable monkeypox viral load (Ct) in oropharyngeal swabs (Number of days)
Viral clearance in rectum swabs | From day 1 to day 57
  Time to undetectable monkeypox viral load (Ct) in rectum swabs (Number of days)
Viral clearance in semen discharge | From day 1 to day 57
  Time to undetectable monkeypox viral load in semen (Number of days)
Viral clearance in vaginal discharge | From day 1 to day 57
  Time to undetectable monkeypox viral load in vaginal discharge (Number of days)

SECONDARY OUTCOMES:
Humoral responses against monkeypox | At baseline and 1, 3, and 6 months later
  Neutralization titers against monkeypox in a subset of participants (Neutralization titers)
Cellular responses against monkeypox | At baseline and 1, 3, and 6 months later
  Presence of specific immunity cells against monkeypox (Presence of cells)

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Atenció Primària Metropolitana Nord, Sabadell, Barcelona
  - Drassanes Vall d'Hebron Centre for International Health and Infectious diseases, Barcelona
  - BCN Checkpoint, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid